CLINICAL TRIAL: NCT03923218
Title: Evaluation of Gingival Crevicular Fluid Levels of LL-37 and Serum Vitamin D3 Levels in Smoker and Non-Smoker Patients With Chronic Periodontitis
Brief Title: Effects of Smoking and Vitamin D3 on the Levels of Human Cathelicidin Peptide LL-37
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gülay Tüter, Professor, Gazi University
Other Study IDs: 03/2011-27
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Periodontitis
Keywords: Gingival crevicular fluid; Vitamin D; LL-37; Serum; periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smoker patients with chronic periodontitis: Smoker patients with chronic periodontitis
  Interventions: Other: LL-37 levels in Gingival crevicular fluid; Other: Serum Vitamin D3 levels; Other: Clinical parameters
- non-smoker patients with chronic periodontitis: non-smoker patients with chronic periodontitis
  Interventions: Other: LL-37 levels in Gingival crevicular fluid; Other: Serum Vitamin D3 levels; Other: Clinical parameters
- periodontally healthy patients: periodontally healthy patients
  Interventions: Other: LL-37 levels in Gingival crevicular fluid; Other: Serum Vitamin D3 levels; Other: Clinical parameters

INTERVENTIONS:
Other: LL-37 levels in Gingival crevicular fluid — Collected gingival crevicular fluid
Other: Serum Vitamin D3 levels — Collected serum
Other: Clinical parameters — Recorded plague index, gingival index, probing depth, clinical attachment level

SUMMARY:
The aims of our study were 1) to evaluate levels of gingival crevicular fluid( GCF) human cathelicidin peptide LL-37 and serum vitamin D3 in smoker and non-smoker patients with chronic periodontitis(CP) 2) to determine whether any correlation between GCF LL-37 and vitamin D3 serum levels exist and 3) to asses the correlation between clinical parameters and biochemical markers

DETAILED DESCRIPTION:
Background: Cathelicidin LL-37, an antimicrobial peptide, is part of the host innate immune response in the oral cavity. The aims of this study are to evaluate; gingival crevicular fluid (GCF) levels of LL-37, serum vitamin D3 levels and periodontal clinical recordings in smoker and nonsmoker patients with chronic periodontitis (CP).

Methods:

This study consisted a total of 60 volunteers including 20 smoker patients with CP (CP-1 group), 20 non-smoker patients with CP (CP-2 group) and 20 periodontally healthy subjects (CTRL group). Prior to participation, the design and purpose of the research were explained to each subjects, and written informed consent form was obtained from 60 individuals before the study.

The periodontal status of the patients were determined by measuring the probing depth (PD), clinical attachment level (CAL), gingival index (GI), plaque index (PI) All clinical parameters were measured on six sites per tooth from the full-mouth teeth (mesiobuccal, distobuccal,midbuccal, mesiolingual, distolingual and midlingual) using a William's periodontal probe calibrated in millimeters by the same examiner. All samples were obtained on the day following clinical examinations of the individuals. The deepest six pockets site per individual were chosen for collection of GCF across both of the periodontitis groups. Six pocket locations showing a lack of clinical inflammation were also tested to guarantee collection of a sufficient volume of GCF across the CTRL groups.

GCF levels of LL-37 were measured by ELISA and serum levels of vitamin D3 were analysed by High-performance liquid chromatography (HPLC). Statistical analysis were performed.

ELIGIBILITY:
Inclusion Criteria for chronic periodontitis groups:

* Clinical attachment loss ≥ 5mm
* Probing depth ≥5mm
* Bone loss affecting >30% of the existing teeth on clinical and radiographic examination
* gingival index (GI) score> 1

Inclusion criteria for control group:

* full-mouth PD was≤ 3mm,
* Gingival index <1
* there was no indication of Attachment Loss or no radiographic evidence of alveolar bone loss in control group.
* Non-smokers.

Smoking criteria for groups:

* patients smoked more than 10 cigarettes in a day
* smoking for 3 or more years,

Exclusion Criteria:

* systemic condition (diabetes, cardiovascular disease, immunologic disorders, hepatitis, e.g.)
* pregnancy, lactation or menopause term,
* antibiotic treatment or non-steroidal anti-inflammatory medications within the last 3 months before the study,
* non-surgical periodontal treatment during the last 6 months before the study,
* treatment with Vitamin D supplementation before the study

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The volunteers participitating in the study were choosen from among individuals scheduled to undergo either dental treatment or dental check at the Deparment of Perioodontology, Faculty of Dentistry, Gazi University, Ankara, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Serum D3 Vitamin levels | Baseline
  The plasma levels of vitamin D3 were greater in the CP-2 group than in the CP-1 group. But, no statistically significant difference was determined between the CP groups (P>0.05)
Gingival Crevicular fluid(GCF) LL-37 levels | Baseline
  The concentration of LL-37 in GCF was significantly higher in both of the CP groups than in the CTRL group (p<0.001). Although GCF LL-37 concentration levels were greater in the CP-1 group than in the CP-2 group, the difference did not reach the statistical significance between the CP groups (p>0.05).

SECONDARY OUTCOMES:
Plaque index (PI) | Baseline
  The full-mouth and sample sites PI recordings were significantly higher in both CP groups (CP-1 and CP-2) than in the CTRL group (p<0.001).
  were measured on six sites per tooth from the full-mouth teeth
GCF volume | Baseline
  The GCF volume was notably higher in both CP groups than in CTRL group (p<0.001).
gingival index (GI) | Baseline
  The full-mouth and sample sites GI recordings were significantly higher in both CP groups (CP-1 and CP-2) than in the CTRL group (p<0.001).
Probing depth (PD) | Baseline
  The full-mouth and sample sites PD recordings were significantly higher in both CP groups (CP-1 and CP-2) than in the CTRL group (p<0.001).
Clinical attachment level (CAL) | Baseline
  The full-mouth and sample sites CAL recordings were significantly higher in both CP groups (CP-1 and CP-2) than in the CTRL group (p<0.001).

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma BOZKURT DOĞAN, Professor, Principal Investigator — university; Elifcan Kıvrak, PhD, Principal Investigator — university